CLINICAL TRIAL: NCT00794014
Title: Optimal Strategy for Side Branch Stenting in Coronary Bifurcation Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-08-073
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- Conservative strategy (Experimental)
  Interventions: Procedure: Conservative strategy
- Aggressive strategy (Experimental)
  Interventions: Procedure: Aggressive strategy

INTERVENTIONS:
Procedure: Conservative strategy — * Main vessel stenting was performed.
  * Side branch ballooning and kissing ballooning were done if Thrombolysis In Myocardial Infarction (TIMI) flow <3 in the side branch after main vessel stenting in non-left main bifurcation (non-LM) subgroup, and diameter stenosis (DS) >75% in LM subgroup.
  * Side branch stenting was performed if TIMI flow <3 in the Side branch after ballooning in non-LM subgroup, and DS >50% or dissection in the Side branch after ballooning in LM subgroup.
  Arms: Conservative strategy
Procedure: Aggressive strategy — * Main vessel was performed.
  * Side branch ballooning and kissing ballooning were done if DS >75% in the side branch after main vessel stenting in non-LM subgroup, and DS >50% in LM subgroup.
  * Side branch stenting was performed if DS >50% in the side branch after ballooning in non-LM subgroup, and DS >30% or dissection in the side branch after ballooning in LM subgroup.
  Arms: Aggressive strategy

SUMMARY:
The purpose of this study is to establish the optimal strategy for side branch stenting in coronary bifurcation lesion.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the relative efficacy and safety of conservative strategy compared to aggressive strategy for side branch stenting in coronary bifurcation lesion.

ELIGIBILITY:
Inclusion Criteria:

* Parent vessel diameter stenosis > 75%
* Parent vessel diameter stenosis 50% - 75% with angina and/or objective evidence of ischemia in the non-invasive stress test
* The reference diameter of both branches more than 2.3 mm by visual estimation

Exclusion Criteria:

* Cardiogenic shock
* ST-elevation myocardial infarction within 48 hours of symptom onset
* Left ventricular dysfunction (echocardiographic left ventricular ejection fraction < 25%)
* Graft vessels
* Patients who have to receive clopidogrel due to other conditions
* Patients who have to receive warfarin, cilostazol or other antiplatelet therapy
* Hypersensitivity to clopidogrel or aspirin
* Expectant survival less than 1 year
* Women who plan to become pregnant
* Patients with bleeding diathesis (coagulopathy, thrombocytopenia or platelet dysfunction, Gastrointestinal or genitourinary bleeding within the prior 3 months)
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2007-11; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | 12 months
  composite of cardiac death, myocardial infarction, target vessel revascularization

SECONDARY OUTCOMES:
Cardiac death | 12 months
  All deaths were considered cardiac unless a definite non-cardiac cause could be established.
Myocardial infarction (MI) | 12 months
  MI was defined as elevated cardiac enzymes (troponin or MB fraction of creatine kinase, CK-MB) more than the upper limit of the normal value with ischemic symptoms or electrocardiography findings indicative of ischemia that was not related to the index procedure.
Target vessel revascularization (TVR) | 12 months
  TVR was repeat revascularization of the target vessel by PCI or bypass graft surgery.
Target lesion revascularization (TLR) | 12 months
  TLR was defined as repeat PCI of the lesion within 5 mm of stent deployment or bypass graft surgery of the target vessel.
Stent thrombosis | 12 months
  Stent thrombosis was assessed based on the definitions of the Academic Research Consortium as definite, probable, or possible stent thrombosis.
Periprocedural enzyme elevation | during the hospitalization
  Periprocedural enzyme elevation was defined as a rise in CK-MB ≥3 times the upper normal limit after the index procedure.
the incidence of binary angiographic restenosis in the main branch and side branch | 9 months
  as measured by 9-month quantitative coronary analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Song YB, Park TK, Hahn JY, Yang JH, Choi JH, Choi SH, Lee SH, Gwon HC. Optimal Strategy for Provisional Side Branch Intervention in Coronary Bifurcation Lesions: 3-Year Outcomes of the SMART-STRATEGY Randomized Trial. JACC Cardiovasc Interv. 2016 Mar 28;9(6):517-26. doi: 10.1016/j.jcin.2015.11.037. PMID 27013152
- [Derived] Song YB, Hahn JY, Song PS, Yang JH, Choi JH, Choi SH, Lee SH, Gwon HC. Randomized comparison of conservative versus aggressive strategy for provisional side branch intervention in coronary bifurcation lesions: results from the SMART-STRATEGY (Smart Angioplasty Research Team-Optimal Strategy for Side Branch Intervention in Coronary Bifurcation Lesions) randomized trial. JACC Cardiovasc Interv. 2012 Nov;5(11):1133-40. doi: 10.1016/j.jcin.2012.07.010. PMID 23174637
- [Derived] Hahn JY, Song YB, Choi JH, Choi SH, Lee SY, Park HS, Hur SH, Lee S, Han KR, Rha SW, Cho BR, Park JS, Yoon J, Lim DS, Lee SH, Gwon HC; DATE Registry Investigators. Three-month dual antiplatelet therapy after implantation of zotarolimus-eluting stents: the DATE (Duration of Dual Antiplatelet Therapy AfterImplantation of Endeavor Stent) registry. Circ J. 2010 Nov;74(11):2314-21. doi: 10.1253/circj.cj-10-0347. Epub 2010 Oct 2. PMID 20938098